CLINICAL TRIAL: NCT01491126
Title: Single Center Open Prospective Study for the Comparison of Procedural Sequence in Same Day Consecutive Bidirectional Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Dan Carter, Gastroenterologist, Gasteroenterologist, Sheba Medical Center
Other Study IDs: SHEBA-11-8951-DC-CTIL
Record Dates: First submitted 2011-12-11; First posted 2011-12-13 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Bidirectional Endoscopy
Keywords: Gastroscopy; Colonoscopy; Anesthesia; Recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- examinees undergoing bidirectional endoscopy: Study population will include sequential examinees undergoing bidirectional endoscopy, age> 18 years

SUMMARY:
The investigators study aim is to determine whether there is a any advantage in starting with upper or lower endoscopy. The main study objective will be the amount of analgesia needed for sustaining the examinee's comfort during the exams. Secondary endpoints will rate of detection of significant pathologies, total time of procedure, examinee's tolerance, time to recovery and examinee's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18
* Same day bidirectional endoscopy

Exclusion Criteria:

* Prior failed endoscopy.
* Any major complication during previous endoscopy.
* Difficulty in communication with the patients.
* Psychiatric disease or mental retardation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include sequential examinees undergoing bidirectional endoscopy. The decision to perform same day sequential bidirectional endoscopy is of the examinee's caring gastroenterologist, and not part of the study. Only examinees > 18 years will be eligible.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Dose of mephridine and midazolam | 1 year
  Dose of analgestices used in order to achive concious sedation

SECONDARY OUTCOMES:
Time to recovery | 1 year
  Time to full recovery and release after endoscopies
Rate of significant findings | 1 year
  Rate of significant findings: colonoscopy: polyps, carcinoma, inflammation, diverticuli, A-V malformations Upper endoscopy: Barret's esophagus, severe esophagitis, gastritis, peptic ulcer disease, polyps and space occupying lesions

CONTACTS AND LOCATIONS:
Overall Officials: Dan Carter, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel

REFERENCES:
- [Background] Cho JH, Kim JH, Lee YC, Song SY, Lee SK. Comparison of procedural sequences in same-day bidirectional endoscopy without benzodiazepine and propofol sedation: starting at the bottom or the top. J Gastroenterol Hepatol. 2010 May;25(5):899-904. doi: 10.1111/j.1440-1746.2009.06157.x. PMID 20546443
- [Background] Urquhart J, Eisen G, Faigel DO, Mattek N, Holub J, Lieberman DA. A closer look at same-day bidirectional endoscopy. Gastrointest Endosc. 2009 Feb;69(2):271-7. doi: 10.1016/j.gie.2008.04.063. Epub 2008 Aug 23. PMID 18725159
- [Background] Hardwick RH, Armstrong CP. Synchronous upper and lower gastrointestinal endoscopy is an effective method of investigating iron-deficiency anaemia. Br J Surg. 1997 Dec;84(12):1725-8. PMID 9448626